CLINICAL TRIAL: NCT04561544
Title: Pilot Test of a Cultural Intervention to Enhance Alaska Native Students' Behavioral Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alaska Anchorage (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Sara Buckingham, Assistant Professor of Psychology, University of Alaska Anchorage
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 1210302; U54GM115371 (NIH)
Record Dates: First submitted 2020-08-30; First posted 2020-09-23 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Depression; Anxiety; Suicidal Ideation; Substance Use
Keywords: Cultural Identity; Sense of Community; Wellbeing; Alaska Native
MeSH Terms: conditions — Depression; Anxiety Disorders; Suicidal Ideation; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention in Fall 2020 (Experimental): Participants will receive the intervention in Fall 2020
  Interventions: Behavioral: Knowing Who You Are (Becoming): Cultural Identity Intervention
- Intervention in Spring 2021 (Other): Control in Fall 2020
  Interventions: Behavioral: Knowing Who You Are (Becoming): Cultural Identity Intervention

INTERVENTIONS:
Behavioral: Knowing Who You Are (Becoming): Cultural Identity Intervention — 8-week cultural identity development program led by Alaska Native Elders

SUMMARY:
This project aims to enhance AN university students' behavioral health by supporting their cultural identity development. While the connection between cultural identity and behavioral health is becoming clearer, comparably less research has explored methods of enhancing identity development. Consequently, the investigators will pilot a cultural identity development program for AN students at the University of Alaska Anchorage (UAA). This intervention is based on extant scientific literature, local findings from focus group with AN students, and traditional wisdom from AN Elders. The eight-week Elder-facilitated program incorporates storytelling, experiential learning, connection, exploration, and sharing of identity, cultural strengths, life paths, and rootedness in who they are in order to remain grounded when they face changes and challenges. Approximately 40 to 50 AN university students will be recruited for the intervention. Participants will be randomized, with half the participants receiving the intervention in the Fall 2020 semester and half the students receiving the intervention in the Spring 2021 semester. We hypothesize that engaging in this intervention will strengthen AN students' cultural identities, strengths, and sense of community; improve their behavioral health, as evidenced in higher self-reported wellbeing, and lower substance use, depression, anxiety, and suicidal ideation symptoms; and support their academic persistence and achievement. Outcomes will be tested via mixed design analyses of covariance. Moreover, program feasibility will be examined through a process evaluation, which will entail thematic analyses of six focus groups with program participants (n=40-50) and with the Elders who facilitated the program (n=5).

ELIGIBILITY:
Inclusion Criteria:

* self-identify as Alaska Native,
* are registered as an undergraduate student at UAA,
* are at least 18 years old,
* speak English

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-08-30 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Degree of Identification with Cultural Identity at Baseline | Baseline, Pre-Intervention
  Multigroup Ethnic Identity Measure (Roberts et al., 1999), a 12-item self-report measure developed for diverse groups that has been validated with Native people (e.g., Moran et al., 1999) to measure cultural identity. Range = 6-30, higher scores indicate greater identification with cultural identity
Change in Baseline Degree of Identification with Cultural Identity Immediately Following Intervention | Immediately After Intervention
  Multigroup Ethnic Identity Measure (Roberts et al., 1999), a 12-item self-report measure developed for diverse groups that has been validated with Native people (e.g., Moran et al., 1999) to measure cultural identity. Range = 6-30, higher scores indicate greater identification with cultural identity
Change in Post-Intervention Degree of Identification with Cultural Identity at 6-Month Follow-Up | Follow-Up, Approximately 6 Months After Intervention
  Multigroup Ethnic Identity Measure (Roberts et al., 1999), a 12-item self-report measure developed for diverse groups that has been validated with Native people (e.g., Moran et al., 1999) to measure cultural identity. Range = 6-30, higher scores indicate greater identification with cultural identity
Degree of Identification with Cultural Strengths at Baseline | Baseline, Pre-Intervention
  Native Cultural Health Assessment Tool (White Shield, 2013), a 10-item self-report measure of cultural strengths in given time period (past month for project) that was developed for Native people to measure cultural strengths. Range = 10-50, higher scores indicate greater identification with cultural strengths.
Change in Baseline Degree of Identification with Cultural Strengths Immediately Following Intervention | Immediately After Intervention
  Native Cultural Health Assessment Tool (White Shield, 2013), a 10-item self-report measure of cultural strengths in given time period (past month for project) that was developed for Native people to measure cultural strengths. Range = 10-50, higher scores indicate greater identification with cultural strengths.
Change in Post-Intervention Degree of Identification with Cultural Strengths at 6-Month Follow-Up | Follow-Up, Approximately 6 Months After Intervention
  Native Cultural Health Assessment Tool (White Shield, 2013), a 10-item self-report measure of cultural strengths in given time period (past month for project) that was developed for Native people to measure cultural strengths. Range = 10-50, higher scores indicate greater identification with cultural strengths.
Strength of Sense of Community with Alaska Native People at University at Baseline | Baseline, Pre-Intervention
  Sense of Community Index, Second Edition (Chavis et al., 2008), a 24-item self-report measure of membership in, shared emotional connection with, fulfillment of needs from, and mutual influence on a given community (e.g., Alaska Native community at UAA) that has been used with diverse populations. Range = 0-72, higher scores indicate greater sense of community.
Change in Baseline Strength of Sense of Community with Alaska Native People at University Immediately Following Intervention | Immediately After Intervention
  Sense of Community Index, Second Edition (Chavis et al., 2008), a 24-item self-report measure of membership in, shared emotional connection with, fulfillment of needs from, and mutual influence on a given community (e.g., Alaska Native community at UAA) that has been used with diverse populations. Range = 0-72, higher scores indicate greater sense of community.
Change in Post-Intervention Strength of Sense of Community with Alaska Native People at University at 6-Month Follow-Up | Follow-Up, Approximately 6 Months After Intervention
  Sense of Community Index, Second Edition (Chavis et al., 2008), a 24-item self-report measure of membership in, shared emotional connection with, fulfillment of needs from, and mutual influence on a given community (e.g., Alaska Native community at UAA) that has been used with diverse populations. Range = 0-72, higher scores indicate greater sense of community.
Degree of Wellbeing at Baseline | Baseline, Pre-Intervention
  Wellbeing scale of the Mental Health Inventory (Veit & Ware, 1983). Converted scores range from 0-100, higher scores indicate greater wellbeing.
Change in Baseline Degree of Wellbeing Immediately Following Intervention | Immediately After Intervention
  Wellbeing scale of the Mental Health Inventory (Veit & Ware, 1983). Converted scores range from 0-100, higher scores indicate greater wellbeing.
Change in Post-Intervention Degree of Wellbeing at 6-Month Follow-Up | Follow-Up, Approximately 6 Months After Intervention
  Wellbeing scale of the Mental Health Inventory (Veit & Ware, 1983). Converted scores range from 0-100, higher scores indicate greater wellbeing.
Degree of Anxiety Symptoms at Baseline | Baseline, Pre-Intervention
  Anxiety scale of the Mental Health Inventory (Veit & Ware, 1983). Converted scores range from 0-100, higher scores indicate more anxiety.
Change in Baseline Degree of Anxiety Symptoms Immediately Following Intervention | Immediately After Intervention
  Anxiety scale of the Mental Health Inventory (Veit & Ware, 1983). Converted scores range from 0-100, higher scores indicate more anxiety.
Change in Post-Intervention Degree of Anxiety Symptoms at 6-Month Follow-Up | Follow-Up, Approximately 6 Months After Intervention
  Anxiety scale of the Mental Health Inventory (Veit & Ware, 1983). Converted scores range from 0-100, higher scores indicate more anxiety.
Degree of Depression Symptoms at Baseline | Baseline, Pre-Intervention
  Depression scale of the Mental Health Inventory (Veit & Ware, 1983). Converted scores range from 0-100, higher scores indicate more depression.
Change in Baseline Degree of Depression Symptoms Immediately Following Intervention | Immediately After Intervention
  Depression scale of the Mental Health Inventory (Veit & Ware, 1983). Converted scores range from 0-100, higher scores indicate more depression.
Change in Post-Intervention Degree of Depression Symptoms at 6-Month Follow-Up | Follow-Up, Approximately 6 Months After Intervention
  Depression scale of the Mental Health Inventory (Veit & Ware, 1983). Converted scores range from 0-100, higher scores indicate more depression.
Degree of Suicidality Symptoms at Baseline | Baseline, Pre-Intervention
  Suicidality scale of the Mental Health Inventory (Veit & Ware, 1983). Converted scores range from 0-100, higher scores indicate more suicidality.
Change in Baseline Degree of Suicidality Symptoms Immediately Following Intervention | Immediately After Intervention
  Suicidality scale of the Mental Health Inventory (Veit & Ware, 1983). Converted scores range from 0-100, higher scores indicate more suicidality.
Change in Post-Intervention Degree of Suicidality Symptoms at 6-Month Follow-Up | Follow-Up, Approximately 6 Months After Intervention
  Suicidality scale of the Mental Health Inventory (Veit & Ware, 1983). Converted scores range from 0-100, higher scores indicate more suicidality.
Degree of Substance Use at Baseline | Baseline, Pre-Intervention
  Items from the Monitoring the Future Survey (U. Michigan), a 9-item self-report measure of tobacco, alcohol, cannabis, cocaine, amphetamine-type stimulants, inhalants, sedatives, hallucinogens, and opioid use in past 30 days. Higher scores indicate greater substance use.
Change in Baseline Degree of Substance Use Immediately Following Intervention | Immediately After Intervention
  Items from the Monitoring the Future Survey (U. Michigan), a 9-item self-report measure of tobacco, alcohol, cannabis, cocaine, amphetamine-type stimulants, inhalants, sedatives, hallucinogens, and opioid use in past 30 days. Higher scores indicate greater substance use.
Change in Post-Intervention Degree of Substance Use at 6-Month Follow-Up | Follow-Up, Approximately 6 Months After Intervention
  Items from the Monitoring the Future Survey (U. Michigan), a 9-item self-report measure of tobacco, alcohol, cannabis, cocaine, amphetamine-type stimulants, inhalants, sedatives, hallucinogens, and opioid use in past 30 days. Higher scores indicate greater substance use.

SECONDARY OUTCOMES:
Academic Achievement at Baseline | Baseline, Pre-Intervention
  Grade point average (GPA) for a given semester.
Change in Baseline Academic Achievement Immediately Following Intervention | Immediately After Intervention
  Grade point average (GPA) for a given semester.
Change in Post-Intervention Academic Achievement at 1-Year Follow-Up | Follow-Up, Approximately 12 Months After Intervention
  Grade point average (GPA) for a given semester.
Rate of Students Maintaining University Enrollment Semester of Intervention | Immediately After Intervention
  Enrollment for a given semester.
Rate of Students Maintaining University Enrollment Semester after Intervention | Follow-Up, Approximately 6 Months After Intervention
  Enrollment for a given semester.
Rate of Students Maintaining University Enrollment One Year Post-Intervention | Follow-Up, Approximately 12 Months After Intervention
  Enrollment for a given semester.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alaska Anchorage, Anchorage, Alaska, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/44/NCT04561544/ICF_000.pdf